CLINICAL TRIAL: NCT03594500
Title: Hearing Impairment, Strategies, and Outcomes in Emergency Departments
Acronym: Hear-VA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 17-068; HX002421-01 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss; Emergency Service; Hospital Readmission
Keywords: Emergency service; Hearing loss; Patient readmission; Communication
MeSH Terms: conditions — Hearing Loss; Communication

STUDY DESIGN:
Intervention Model Description: Consenting participants will be randomly assigned to the control or intervention arm of the study. Participants in the intervention arm will receive PockeTalkers (hearing assistance devices) for the duration of their time in the emergency department. Participants in the control group will not receive hearing assistance devices during their time in the emergency department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: PockeTalker (Experimental): Consenting participants will be randomly assigned to the intervention group while receiving care in the emergency department
  Interventions: Other: PockeTalker
- Control: No PockeTalker (Other): Consenting participants will be randomly assigned to the control group while receiving care in the emergency department
  Interventions: Other: No PockeTalker

INTERVENTIONS:
Other: PockeTalker — The intervention group will receive PockeTalkers (hearing assistance devices) while they receive care in the ED
  Other Names: Hearing Assistance Device
  Arms: Intervention: PockeTalker
Other: No PockeTalker — The control group will not receive PockeTalkers while they receive care in the ED
  Arms: Control: No PockeTalker

SUMMARY:
Aim 1: Establish the feasibility of screening for hearing loss in the ED Aim 2: Determine the acceptability of the screening procedure (among the ED population) Aim 3: Derive a preliminary estimate of the effect size of primary outcomes Aim 4: Identify the evidence that decision makers in Veteran Affair Medical Centers, ED and Audiology Services need to commit to this approach

DETAILED DESCRIPTION:
The goal of this study is to test whether providing hearing assistance devices to older age hearing impaired patients in the ED setting will improve in-ED understanding and preparation for discharge. The proposed intervention, the Hearing Impairment, Strategies and Outcomes in VA Emergency Departments (HearVA-ED) will be conducted in the Emergency Departments of the Manhattan and Brooklyn VAs of the New York Harbor Healthcare System and will recruit hearing impaired ED patients who are 60 years and older and have been admitted to the ED with a low acuity triage score indicating a high likelihood of discharge home. The investigators will identify hearing impairment by using the Hearing Handicap Inventory for the Elderly survey (HHIE-S). The investigators will randomize consenting patients who fail the screening to either receipt of a simple hearing assistance device (a "PockeTalkerTM") during their ED stay or usual care. The investigators will test whether the provision of a PockeTalkerTM is feasible in this environment (by measuring the amount of device use), whether providing the device improves self-reported quality of hearing and understanding during the ED stay, and whether use of the device improves the quality of preparation for post-discharge care. If this randomized controlled trial demonstrates beneficial effects for in-ED use of a simple hearing assistance device for hearing impaired patients, this strategy can be disseminated throughout the VA healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Emergency severity index criterion of 4 or 5 (low acuity)
* Hearing Handicap Impairment Evaluation Screen greater than or equal to 24
* Capacity to consent to participate in research

Exclusion Criteria:

* Inability to consent to participate in research
* Emergency severity index criterion of 1-3 (high acuity)
* Hearing Handicap Impairment Evaluation Screen less than 24
* Inability to speak English or Spanish

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD MSHS, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Started | 66 | 67
Completed | 60 | 63
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: The first phase of intervention, the Hearing Impairment, Strategies and Outcomes in VA Emergency Departments (HearVA-ED) was conducted in the Emergency Departments of the Manhattan and Brooklyn VAs of the New York Harbor Healthcare System and recruited hearing impaired ED patients who are 60 years and older and were admitted to the ED with a low acuity triage score indicating a high likelihood of discharge home.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 56 | 62 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (9.36) | 76.2 (9.09) | 76.4 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 65 | 65 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 20
  Not Hispanic or Latino | 50 | 61 | 111
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 43 | 44 | 87
  Race/Ethnicity: Black | 19 | 19 | 38
  Race/Ethnicity: Asian | 1 | 1 | 2
  Race/Ethnicity: Unknown/Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 67 | 133
Education Level [Count of Participants; unit: Participants]
  Less than high school | 4 | 5 | 9
  Completed high school | 12 | 15 | 27
  Some college | 17 | 14 | 31
  Completed college | 30 | 28 | 58
  Missing | 3 | 5 | 8
Primary Language [Count of Participants; unit: Participants]
  English | 46 | 57 | 103
  Spanish | 5 | 1 | 6
  Other | 12 | 4 | 16
  Missing | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Use of Hearing Assistance Device (HAD) During Emergency Department (ED) Stay
Description: The investigators will observe and survey intervention participants to determine whether or not they use the hearing assistance device while they are in the ED. This will be measured on a yes/no basis.
Time Frame: Duration of ED stay, average of 1-2 days
Population: Those randomized to receive the hearing assistance device, how many used the hearing assistance device in the ED
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: received hearing assistance device: (randomized to receive hearing assistance device)
Arm/Group | Intervention: received hearing assistance device
Number analyzed (Participants) | 63
Participants
  Yes (Used a hearing assistance device) | 38
  No (Did not use a hearing assistance device) | 25

2. Primary Outcome: Patient-Rated Quality of Hearing, Understanding, and Communication With Providers During ED Stay
Description: Participants will self-rate their quality of hearing, understanding, and communication using a six item questionnaire. Scored on a 10-point Likert scale (1 = do not agree at all; 10 = completely agree) the questions will be: When I talked to the doctors and nurses today ... (1) their voices were very clear; (2) I was able to hear the sounds that I wanted to hear; (3) noises did not cause a problem for my hearing; and (4) listening did not make me tired. Two additional statements will explicitly capture understanding: (5) I was able to understand what they said; and (6) I was able to understand without making an effort. Higher scores will indicate better communication and understanding with providers.
Time Frame: Duration of ED stay, average of 1-2 days
Measure: Number; unit: Percent of participants
Groups:
- Intervention: Veterans who received HAD in ED
- Control: Veterans who did not receive HAD in ED
Arm/Group | Intervention | Control
Number analyzed (Participants) | 60 | 63
Percent of participants
  1. Their voices were very clear. | 90 | 84
  2. I was able to hear the sounds that I wanted to hear. | 81 | 79
  3. Noises did not cause a problem for my hearing. | 69 | 66
  4. Listening did not make me tired. | 89 | 74
  5. I was able to understand what they said. | 90 | 84
  6. I was able to understand without making an effort. | 76 | 56

3. Primary Outcome: Patient-Rated Quality of Post-Discharge Care
Description: Patient-rated quality of post-discharge care using a three-item subset of the Care Transition Measure (CTM). The questions are scored on a 1-4 scale (1= strongly disagree; 4 = strongly agree): (1) The ED staff considered my preferences and those of my family or caregiver in deciding what my healthcare needs were for discharge; (2) Leaving the ED, I have a good understanding of the things I am responsible for in managing my health; (3) Leaving the ED, I clearly understand the purpose for each of my medications. Higher scores will indicate better discharge preparation.
Time Frame: At time of discharge from ED, average 1 day
Measure: Number; unit: percentage of participants who agree
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 60 | 63
percentage of participants who agree
  1. ED staff took my preferences into account in deciding my health care needs when I left. | 95 | 90
  2. I have a good understanding of my responsibilities for managing my health. | 97 | 85
  3. When leaving, I clearly understood the purpose for taking each of my medications. | 97 | 93

4. Secondary Outcome: Education Level
Description: The Investigators will code what education level the Veterans have completed.
Time Frame: Duration of ED stay, average of 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 63 | 62
Participants
  Education: Less than high school | 4 | 5
  Education: Completed high school | 12 | 15
  Education: Completed college | 30 | 28
  Education: Some college | 17 | 14

5. Secondary Outcome: Primary Language
Description: The Investigators will code what language the Veterans speak when at home.
Time Frame: Duration of ED stay, average of 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 63 | 62
Participants
  English | 46 | 57
  Spanish | 5 | 1
  Other | 12 | 4

6. Secondary Outcome: Number of Participants Who Live Alone or With Others
Description: The Investigators will code whether the Veteran lives with others or alone.
Time Frame: Duration of ED stay, average of 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 63 | 62
Participants
  Yes (Lives Alone) | 34 | 43
  No (Lives with Others) | 29 | 19

7. Secondary Outcome: Number of Participants in the ED Alone or With Others
Description: The Investigators will code whether the Veteran came to the ED with others or alone.
Time Frame: Duration of ED stay, average of 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 66 | 67
Participants
  Yes (At ED Alone) | 45 | 55
  No (At ED with Others) | 21 | 12

8. Secondary Outcome: Hospital Readmission
Description: The Investigators will determine whether patients have had an ED revisit within three and 30 days through CPRS review as well as a brief follow-up phone call four and 35 days after ED discharge.
Time Frame: 3-30 days after initial ED stay
Population: The Investigators will determine whether patients have had an ED revisit within three and 30 days through CPRS review as well as a brief follow-up phone call four and 35 days after ED discharge at the conclusion of phase 2 of the project.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention: PockeTalker | Control: No PockeTalker
Number analyzed (Participants) | 60 | 63
percentage of participants
  3-day readmissions | 3 | 9
  30-day readmissions | 23 | 27

ADVERSE EVENTS:
Time Frame: 35 days post-discharge
Description: The definition of an adverse event and/or serious adverse event, used to collect adverse event information does not differ from the clinical trial definitions.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/67
Other Adverse Events (participants affected / at risk) | 0/66 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT03594500/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03594500/SAP_001.pdf